CLINICAL TRIAL: NCT05288387
Title: Hemodynamic Effects of Transcutaneous Spinal Cord Stimulation in Patients With Chronic Heart Failure Undergoing Right Heart Catheterization for the Inclusion Into the Heart Transplantation Program: a Pilot Study
Brief Title: Spinal Cord Stimulation in Hypotensive Heart Failure Patients: Hemodynamic Assessment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No perceivable effect of transcutaneous spinal cord stimulation on blood pressure in heart failure patients
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HF-SCS-2022
Record Dates: First submitted 2022-01-28; First posted 2022-03-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation in heart failure patients with hypotension (Experimental): Adhesive patches are applied to subjects' back skin. Single stimuli are delivered in order to define the stimulation threshold under the guidance of neuromyography. Vascular access is performed (jugular or subclavian) according to conventional preparation to right heart catheterization. Invasive hemodynamic measures are performed as usual.
  High-frequency spinal cord stimulation at T5 level is initiated, and repeated hemodynamic measures performed within 2 minutes. Stimulation lasts for 5-10 minutes, and then ceased. Following a 5-minutes waiting period, repeat hemodynamic measures are performed. The same sequence of steps applies for stimulation levels T7-8 and a combination of T5 and T7-8.
  Then the procedure is completed and data are analysed.
  Interventions: Procedure: Spinal cord stimulation

INTERVENTIONS:
Procedure: Spinal cord stimulation — High-frequency stimulation with modulated current via skin patches captures posterior horns of the spinal cord and this activation leads to blood pressure elevation.

SUMMARY:
This is a prospective single-center study that aims to evaluate the effects of non-invasive transcutaneous spinal cord stimulation on systemic and pulmonary hemodynamics, assessed during right heart catheterization in patients with heart failure and persistent or transient hypotension subjected to be included into the heart transplantation waiting list.

DETAILED DESCRIPTION:
The study aims to assess hemodynamic effects of non-invasive transcutaneous spinal cord stimulation during invasive hemodynamics evaluation in patients with heart failure and transient or persistent hypotension undergoing catheterization before inclusion into the heart transplantation program. Eligible patients will sign an informed consent form before the procedure. Non-invasive transcutaneous electrical stimulation of the spinal cord will be applied using high-frequency modulated electrical impulses through adhesive electrodes attached to the back skin. The stimulation protocol includes analysis of the following parameters: heart rate; electrocardiogram in 12 leads; invasive blood pressure; pulmonary artery pressure, pulmonary capillary wedge pressure, cardiac input, cardiac index, stroke volume, stroke volume index, systemic vascular resistance, pulmonary vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Patients with heart failure III-IV functional class (NYHA) with indications to right heart catheterization.
3. Systolic blood pressure <110/70 mm Hg when measured while sitting.
4. Patient who signed an informed consent form.

Exclusion Criteria:

1. Hypovolemic status (central venous pressure <2 mm Hg).
2. Any acute illness.
3. Transient ischemic event or stroke within 2 weeks prior to inclusion.
4. Pulmonary embolism <1 month ago.
5. Epilepsy.
6. An implanted infusion pump.
7. Pacemaker-dependent patients.
8. Patients who have contraindications to the use of the patch electrodes used in this study, as indicated in the respective instructions for use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure elevation | 10 minutes
  It is suggested that spinal cord stimulation will elevate averaged systolic blood pressure by >5 mmHg within 10 minutes, as compared to tilt testing without stimulation, and as measured invasively through a vascular catheter. Number of participants with increase in systolic blood pressure by more than 5 mmHg within 10 minutes will be counted. The achievement of the primary outcome will be considered if >50% of patients will have an increase in systolic blood pressure.

SECONDARY OUTCOMES:
Systemic vascular resistance elevation | 10 minutes
  It is suggested that spinal cord stimulation will elevate systemic vascular resistance by 10 percent (estimated using the standard equation method based on invasive hemodynamic measurements). Hemodynamic measures are performed using a hemodynamic catheter. This is a physiological parameter. Number of patients with change >10 percent will be calculated.
Pulmonary vascular resistance change | 10 minutes
  A statistically detectable decrease in pulmonary vascular resistance in the patient group based on invasive hemodynamic measurements, and estimated using the standard equation method based on invasive hemodynamic measurements. Hemodynamic measures are performed using a hemodynamic catheter. This is a physiological parameter. Number of patients with change >10 percent will be calculated.
Pulmonary capillary wedge pressure change | 10 minutes
  A statistically detectable change in pulmonary capillary wedge pressure in the patient group based on invasive measurements. Hemodynamic measures are performed using a hemodynamic catheter. This is a physiological parameter. Number of patients with change >10 percent will be calculated.
Pulmonary artery pressure change | 10 minutes
  A statistically detectable change in pulmonary artery systolic, diastolic, or mean pressure in the patient group based on invasive measurements. Hemodynamic measures are performed using a hemodynamic catheter. This is a physiological parameter. Number of patients with change >10 percent will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny N Mikhaylov, Assoc.prof., Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed during regular meetings of the study and supervising committees after enrollment of at least 30% of subjects.

REFERENCES:
- [Background] Mikhaylov EN, Moshonkina TR, Zharova EN, Garkina SV, Kovzelev PD, Belyaeva NN, Kozlenok AV, Lebedev DS, Shlyakhto EV. Acute Cardiovascular Effects of Non-Invasive Electrical Spinal Cord Stimulation: Results from a Pilot Study in Humans. J Cardiovasc Transl Res. 2020 Dec;13(6):891-893. doi: 10.1007/s12265-020-10014-7. Epub 2020 May 6. PMID 32378161